CLINICAL TRIAL: NCT00471250
Title: Research Respiratory Tract Procedures
Brief Title: Collection of Lung Fluid and Tissue Samples for Research
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070142; 07-H-0142
Record Dates: First submitted 2007-05-08; First posted 2007-05-09 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-12-18

CONDITIONS: Leukocyte Disorders; Respiratory Tract Diseases; Bronchoscopy
Keywords: Lung Infection Susceptibility; Bronchoalvealar lavage; Nasal Biopsy; Sputum Sample; Infection Susceptibility; Natural History; Healthy Volunteer; HV
MeSH Terms: conditions — Leukocyte Disorders; Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Healthy Volunteers
- 2: NIH patients with known or suspected susceptibility to infection.

SUMMARY:
This study will collect fluid and tissue specimens from the lungs and nose of healthy people and people with a history of lung infections. The specimens will be examined for differences between the two groups that may be associated with susceptibility to certain infections.

Healthy normal volunteers and people with a history of lung infections between 18 and 75 years of age who are followed at NIH may be eligible for this study.

Participants undergo the following procedures:

Medical history and physical examination.

Blood and urine tests.

Electrocardiogram (ECG) and chest x-ray.

Treadmill exercise stress test (for people over 45 years old with a history of chest pain or ECG abnormalities).

Bronchoscopy: The subject s nose and throat are numbed with lidocaine and a sedative is given for comfort. A thin flexible tube called a bronchoscope is advanced through the nose or mouth into the lung airways to examine the airways carefully.

Fluid collection during the bronchoscopy using one of the following methods:

* Bronchoalveolar lavage: Salt water is injected through the bronchoscope into the lung and immediately suctioned out, washing off cells lining the airways.
* Bronchial brushings: A brush-tipped wire enclosed in a sheath is passed through the bronchoscope and a small area of the airway tissue is gently brushed. The brush is withdrawn with some tissue adhering to it.
* Endobronchial biopsies: Small pinchers on a wire are passed through the bronchoscope and about 1 to 2 millimeters of tissue is removed.
* Nasal scrape: A small device is used to scrape along the inside of the nose to collect some cells.
* Sputum induction
* Exhaled breath condensate to obtain specimens for in vitro investigations and comparisons of both the cellular and acellular components.
* Nasal nitric oxide production
* Nasal potential difference
* Exhaled aerosol mask sample collection
* Cough aerosol collection
* Exhaled particle collection
* Lung Clearance Index (LCI)

DETAILED DESCRIPTION:
This research protocol involves one or more of the following procedures in healthy volunteers and patients with known or suspected predisposition to respiratory infection who are enrolled in National Institutes of Health (NIH) protocols: 1) Adults only: bronchoscopy with sampling of bronchoalveolar lavage fluid and epithelial cells in healthy adult volunteers and patients; 2) Adults and Children: sputum induction for collection of sputum specimens; 3) Adults and Children: nasal mucosal biopsies and brushings for sampling of epithelial cells; 4) Adults and Children: measurement of nasal nitric oxide production; 5) Adults and children: collection of exhaled breath condensate; 6) Adults and children: measurement of nasal potential difference; 7) Adults and children: exhaled aerosol mask sample collection; Adults and children: 8) cough aerosol collection. The cellular and acellular samples will be separated, and stored or transferred to the appropriate laboratories investigating these diseases.

Alveolar macrophages are the predominant (>95%) cell type present in the lavage of normal subjects. Alveolar macrophages play a central role in the initiation and propagation of lung inflammation by releasing cytokines (i.e., interleukin-1, tumor necrosis factor) and chemokines (i.e., interleukin-8, monocyte chemotactic protein, macrophage inflammatory protein) that activate other resident cells and recruit inflammatory cells to a local nidus of inflammation. Airway epithelial cells are known to release a variety of mediators as well. Thus, the interaction of cells with mediators generated by alveolar cells and bronchial epithelial cells during acute inflammation is a key element in the initiation of pulmonary inflammatory responses.

Bronchoalveolar lavage (BAL), bronchial brushings, and mucosal biopsies are standard diagnostic techniques done through the bronchoscope to obtain samples of alveolar and bronchial specimens for diagnosis of infection, malignancy, or non-infectious inflammation. Nasal mucosal scrape biopsy is a minimally invasive method of obtaining airway epithelial cells to diagnose disorders of airway clearance associated with abnormal cilia (hair-like structures on airway lining cells). Sputum induction is a routinely performed procedure to facilitate the collection of respiratory secretions (mucus) through stimulation of cough with inhalation of an aerosolized concentrated salt-water solution. Exhaled breath condensate is simply collected by breathing normally through a plastic tube inserted into a chilled cylinder. Nasal potential difference is performed by placing a small needle under the skin of the forearm that is connected to a salt solution bridge and resting a small catheter on the surface of the nose through which various salt solutions are dripped.

The objective of this protocol is to analyze bronchoalveolar lavage fluid, airway epithelial cells, sputum, and exhaled breath specimens and bedside physiologic measurements from healthy volunteers and from patients who acquire respiratory infections to look for differences in immune function and to discover new pathways of infectious disease susceptibility. We hypothesize that studying cellular responses to infection and inflammatory markers released from these cells will further our understanding of human susceptibility to respiratory tract infections.

Five hundred fifty subjects (250 healthy volunteers and 300 patients) will undergo one or more of the following: 1) bronchoscopy with bronchoalveolar lavage, bronchial brushings, endobronchial biopsies; 2) nasal mucosal scrape and/or brush biopsies; 3) sputum induction 4) exhaled breath condensate to obtain specimens for in vitro investigations and comparisons of both the cellular and acellular components. Bedside measurements 5) nasal nitric oxide production and 6) nasal potential difference 7) exhaled aerosol mask sample collection 8) cough aerosol collection 9) Exhaled particle collection; 10) Lung Clearance Index

(LCI) may be done to assess airway infection and epithelial cell functions in real-time.

ELIGIBILITY:
* HEALTHY VOLUNTEER INCLUSION CRITERIA FOR BRONCHOSCOPY AND BRONCHOSCOPIC PROCEDURES:

  1. 18 to 75 years of age inclusive
  2. Enrolled without regard to gender, race, or ethnicity
  3. NIH staff are eligible
  4. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
  5. Able and willing to complete the informed consent process
  6. Able and willing to arrange to have another person drive them home after the procedure
  7. Able and willing not to eat or drink anything for 6 hours prior and 2 hours after the procedure
  8. Willing to donate blood and respiratory tract samples for storage to be used for future research
  9. In good general health without clinically significant medical history
  10. Physical examination without clinically significant findings
  11. Screening laboratory tests without clinically significant abnormalities:
* Complete blood count with differential
* Serum chemistries including creatinine, blood urea nitrogen, glucose, liver enzymes and function tests, electrolytes
* HIV test and hepatitis serologies (HBsAg; HCV) if status is unknown
* Prothrombin time, partial thromboplastin time
* Urinalysis
* Female subjects must have negative urine pregnancy test within 1 week of participation and continue birth control practices prior to participation
* Chest radiograph (CXR) (if the subject has not had a CXR or computerized tomography [CT] scan of the chest within the prior 7 days)
* Pulse oximetry
* Electrocardiogram (ECG)
* Treadmill exercise stress test (as indicated for history of angina or abnormalities on ECG)

HEALTHY VOLUNTEER EXCLUSION CRITERIA FOR BRONCHOSCOPY AND BRONCHOSCOPIC PROCEDURES:

1. <18 or >75 years old
2. A smoking history of 10 pack-years or more, a current smoker, or tobacco free for less than a year.
3. Positive HIV status. Subjects must have a negative FDA-approved HIV blood test. [Note: Results of HIV enzyme-linked immunosorbent assay (ELISA) will be documented, but a negative HIV polymerase chain reaction (PCR) test result will be sufficient for eligibility screening of subjects with positive HIV ELISA that is due to prior participation in an HIV vaccine study]
4. Acute or chronic hepatitis based on viral hepatitis serologies
5. Pregnancy or breastfeeding
6. Any active medical problems especially bleeding disorders, significant bruising or bleeding difficulties with intramuscular (IM) injections or blood draws, use of anticoagulants, or pulmonary disorders including asthma
7. History of allergic reaction to lidocaine, sedative medications like Valium Trademark or Versed Trademark, or narcotic medications like morphine or fentanyl
8. Immunosuppressive medications, cytotoxic medications, inhaled corticosteroids, or long-acting beta-agonists within the past three months. (Note that use of corticosteroid nasal spray for allergic rhinitis, topical corticosteroids for an acute uncomplicated dermatitis, or short-acting beta-agonists in controlled asthmatics is not excluded).
9. Use of platelet inhibitors including aspirin and nonsteroidal anti-inflammatory drugs (NSAIDs) within 7 days of procedure
10. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer s ability to give informed consent

PATIENT INCLUSION CRITERIA FOR BRONCHOSCOPY AND BRONCHOSCOPIC PROCEDURES

1. 18 to 75 years of age inclusive
2. Known or suspected respiratory infections or infection susceptibility
3. Enrolled without regard to gender, race, or ethnicity
4. Must be enrolled in a concurrent NIH protocol and under the care of a primary physician outside of the NIH
5. Able and willing to complete informed consent process
6. Able and willing to arrange to have another person drive them home after the procedure
7. Able and willing not to eat or drink anything for 6 hours prior and 2 hours after the procedure
8. Willing to donate blood and respiratory tract samples for storage to be used for future research

PATIENT EXCLUSION CRITERIA FOR BRONCHOSCOPY AND BRONCHOSCOPIC PROCEDURES

1. <18 or >75 years old
2. History of recent/acute clinically significant pulmonary compromise. This will be defined by the following criteria:

   * New lung infection or change in status of chronic lung infection or significant new findings on chest x-ray or CT scan
   * Asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past two years, or that required the use of oral or parenteral corticosteroids during the past two years
   * Clinically significant reactive airway disease that does not respond to bronchodilators
   * Unstable chronic lung disease such as Chronic Obstructive Pulmonary Disease (COPD) or pulmonary fibrosis
   * History of pulmonary hypertension
   * Requirement of supplemental oxygen at rest
3. Unstable angina or uncontrolled heart failure or rhythm disturbance
4. Significant kidney or liver disease
5. Significant anemia with a hemoglobin of less than 7.5 grams/dl.
6. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions), significant bruising or bleeding difficulties with IM injections or blood draws, or use of anticoagulant medications
7. Use of platelet inhibitors including aspirin and NSAIDs within 7 days of procedure or clopidogrel (Plavix Trademark) within 14 days of procedure or the inability to safely stop platelet inhibitors for 7-14 days prior to procedures
8. History of allergic reaction to lidocaine, sedative medications like Valium Trademark or Versed Trademark, or narcotic medications like morphine or fentanyl
9. Pregnancy or breastfeeding
10. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

HEALTHY VOLUNTEER INCLUSION CRITERIA FOR NASAL MUCOSAL BIOPSY, NASAL NITRIC OXIDE MEASUREMENT, AND NASAL POTENTIAL DIFFERENCE MEASUREMENT:

1. >= 5 years old
2. Enrolled without regard to gender, race, or ethnicity
3. NIH staff are eligible
4. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
5. Able and willing to complete the informed consent process
6. Willing to donate blood and respiratory tract samples for storage to be used for future research
7. Stable vital signs

HEALTHY VOLUNTEER EXCLUSION CRITERIA FOR NASAL MUCOSAL BIOPSY, NASAL NITRIC OXIDE MEASUREMENT, AND NASAL POTENTIAL DIFFERENCE MEASUREMENT:

1. <5 years old
2. History of frequent colds or significant uncontrolled hay fever symptoms, recent or active upper respiratory tract infection, such as a cold or sinusitis, or chronic sinus infection or congestion
3. History of turbinectomy or significant nasal pathology that would preclude obtaining mucosal scrape biopsies or other measures
4. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions), significant bruising or bleeding difficulties with IM injections or blood draws, or use of anticoagulant medications
5. The use of nasal steroids in the past 6 weeks
6. Any medical, psychiatric, social condition, occupational reason, or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer s ability to give informed consent

PATIENT INCLUSION CRITERIA FOR NASAL MUCOSAL BIOPSY, NASAL NITRIC OXIDE MEASUREMENT, NASAL POTENTIAL DIFFERENCE MEASUREMENT, SPUTUM INDUCTION, COUGH AEROSOL SAMPLING, EXHALED AEROSOL MASK SAMPLE COLLECTION, COLLECTION OF EXHALED PARTICLES, AND LCI:

1. >= 5 years old
2. Known or suspected infections or infection susceptibility
3. Enrolled without regard to gender, race, or ethnicity
4. Must be enrolled in a concurrent NIH protocol and under the care of a primary physician outside of the NIH
5. Able and willing to complete informed consent process
6. Willing to donate blood and respiratory tract samples for storage to be used for future research

PATIENT EXCLUSION CRITERIA FOR NASAL MUCOSAL BIOPSY, NASAL NITRIC OXIDE MEASUREMENT, NASAL POTENTIAL DIFFERENCE MEASUREMENT, SPUTUM INDUCTION, COUGH AEROSOL SAMPLING, EXHALED AEROSOL MASK SAMPLE COLLECTION, COLLECTION OF EXHALED PARTICLES, AND LCI:

1. <5 years old
2. Significant uncontrolled hay fever symptoms or recent or active upper respiratory tract infection, such as a cold or sinusitis
3. History of turbinectomy or significant nasal pathology that would preclude obtaining mucosal scrape biopsies or other measures
4. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions), significant bruising or bleeding difficulties with IM injections or blood draws, or use of anticoagulant medications
5. Any medical, psychiatric, social condition, occupational reason, or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

HEALTHY VOLUNTEER INCLUSION CRITERIA FOR SPUTUM INDUCTION, EXHALED BREATH CONDENSATE COLLECTION COUGH AEROSOL SAMPLING, EXHALED AEROSOL MASK SAMPLE COLLECTION, COLLECTION OF EXHALED PARTICLES, AND LCI:

1. >= 5 years old
2. Enrolled without regard to gender, race, or ethnicity
3. NIH employees or non-employees eligible
4. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
5. Able and willing to complete the informed consent process
6. Willing to donate blood and respiratory tract samples for storage to be used for future research
7. Stable vital signs

HEALTHY VOLUNTEER EXCLUSION CRITERIA FOR SPUTUM INDUCTION, EXHALED BREATH CONDENSATE COLLECTION, COUGH AEROSOL SAMPLING, EXHALED AEROSOL MASK SAMPLE COLLECTION, COLLECTION OF EXHALED PARTICLES, AND LCI:

1. < 5 years old
2. History of asthma or reactive airways disease
3. Any medical, psychiatric, social condition, occupational reason, or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer s ability to give informed consent

PATIENT INCLUSION CRITERIA FOR SPUTUM INDUCTION, EXHALED BREATH CONDENSATE COLLECTION, COUGH AEROSOL SAMPLING, EXHALED AEROSOL MASK SAMPLE COLLECTION, COLLECTION OF EXHALED PARTICLES, AND LCI:

1. >= 5 years old
2. Known or suspected infections or infection susceptibility
3. Enrolled without regard to gender, race, or ethnicity
4. Must be enrolled in a concurrent NIH protocol and under the care of a primary physician outside of the NIH
5. Able and willing to complete informed consent process
6. Willing to donate blood and respiratory tract samples for storage to be used for future research

PATIENT EXCLUSION CRITERIA FOR SPUTUM INDUCTION, EXHALED BREATH CONDENSATE, COUGH AEROSOL SAMPLING, EXHALED AEROSOL MASK SAMPLE COLLECTION, COLLECTION OF EXHALED PARTICLES, AND LCI:

1. < 5 years old
2. Significant uncontrolled asthma or reactive airways disease
3. Any medical, psychiatric, social condition, occupational reason, or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer s ability to give informed consent.

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteers and NIH patients with known or suspected susceptibility to infection.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2007-08-17 (Actual)

PRIMARY OUTCOMES:
obtain bronchoalveolar lavage fluid, sputum, and/or airway epithelial cells from healthy volunteers and from patients who acquire respiratory infections, to look for differences in immune function between these groups, and to discover new pat... | 10 years
  to obtain respiratory tract cells fluids, and bedside physiologic measurements from normal and diseased subjects to support current bench research studies or to be stored for future studies.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Lipton, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Busse WW, Wanner A, Adams K, Reynolds HY, Castro M, Chowdhury B, Kraft M, Levine RJ, Peters SP, Sullivan EJ. Investigative bronchoprovocation and bronchoscopy in airway diseases. Am J Respir Crit Care Med. 2005 Oct 1;172(7):807-16. doi: 10.1164/rccm.200407-966WS. Epub 2005 Jul 14. PMID 16020805
- [Background] Goldstein RA, Rohatgi PK, Bergofsky EH, Block ER, Daniele RP, Dantzker DR, Davis GS, Hunninghake GW, King TE Jr, Metzger WJ, et al. Clinical role of bronchoalveolar lavage in adults with pulmonary disease. Am Rev Respir Dis. 1990 Aug;142(2):481-6. doi: 10.1164/ajrccm/142.2.481. PMID 2200319
- [Background] Bush A, Pohunek P. Brush biopsy and mucosal biopsy. Am J Respir Crit Care Med. 2000 Aug;162(2 Pt 2):S18-22. doi: 10.1164/ajrccm.162.supplement_1.maic-5. No abstract available. PMID 10934126
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2007-H-0142.html